CLINICAL TRIAL: NCT00069173
Title: Prevention of Osteoporosis Among Sedentary Adolescent Females
Brief Title: Preventing Osteoporosis in Adolescent Girls
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R01HD037746 (NIH)
Record Dates: First submitted 2003-09-16; First posted 2003-09-17 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-06

CONDITIONS: Osteoporosis
Keywords: Females; Sedentary; School-based
MeSH Terms: conditions — Osteoporosis; Sedentary Behavior

INTERVENTIONS:
Behavioral: Project FAB (Fitness and Bone)

SUMMARY:
Physical activity in adolescents is an important part of bone health. Good bone health in adolescents can decrease the risk of osteoporosis. This study will evaluate a program designed to increase the level of physical activity in adolescent girls.

DETAILED DESCRIPTION:
Despite the documented health benefits of increased physical activity, there is limited research on behavioral programs designed to increase exercise in adolescents. Psychosocial characteristics, such as self-efficacy for exercise, social support for exercise from family and peers, and perceived benefits of and barriers to exercise, may predispose adolescents toward the adoption and maintenance of physical activity. This study will implement a multifaceted behavioral program specifically designed to increase bone strengthening physical activity by addressing many of the psychosocial factors relating to exercise.

Girls in this study will be enrolled in Project Fitness and Bone (FAB). The Project FAB intervention is delivered during a regular school class period 5 days per week for 10 months. One day per week is devoted to didactic presentations and/or discussion about reasons for being active, ways of overcoming barriers to being active, and strategies for maintaining an active lifestyle. The remaining four days are structured activity sessions, including a range of activities such as modified basketball, aerobic dance, and walking around a track. Primary outcome measures will include bone mass (measured via dual-energy x-ray absorptiometer [DEXA]) and serum and urinary measures of bone formation and resorption. Participants will be contacted by telephone 12 months after their final clinic visit to ascertain their activity level at that time.

ELIGIBILITY:
Inclusion Criteria

* Entering the 10th or 11th grade
* Participating in fewer then three vigorous activity sessions per week lasting 20 minutes or more or fewer than five moderate activity sessions per week lasting 30 minutes or more
* At or below the 75 percentile for age- and gender-specific cardiovascular fitness
* Past the age of first menstrual cycle

Exclusion Criteria

* Health problems that would preclude participation in regular exercise

Ages: 13 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 250
Dates: Start 2000-07

CONTACTS AND LOCATIONS:
Overall Officials: Margaret S. Jamner, PhD, Principal Investigator — University of California at Irvine
Locations (1):
- University of California at Irvine, Irvine, California, United States